CLINICAL TRIAL: NCT07070414
Title: Alcohol and Cannabis Use Among Assault-Injured Emerging Adults
Brief Title: Substance Use in Assault-Injured Young Adults
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2000040490; 1R34DA061051-01A1 (NIH)
Record Dates: First submitted 2025-07-08; First posted 2025-07-17 (Actual); Last update posted 2025-11-03 (Actual); Status verified 2025-10

CONDITIONS: Alcohol Misuse; Cannabis Misuse
Keywords: alcohol misuse; cannabis misuse
MeSH Terms: interventions — Acclimatization

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Brief Negotiation Interview intervention (BNI) (adapted) (Experimental): Participants randomized to the intervention arm will receive a brief motivational interview designed to increase motivation to reduce alcohol and/or cannabis use and engagement in treatment referral at 30-days. A referral includes a contact number to addiction treatment (primary care and/or specialty addiction care consistent with diagnostic criteria) and injury prevention services at the Yale Hospital Violence Intervention Program.
  Interventions: Behavioral: Brief Negotiation Interview intervention (BNI) (adapted)
- Control Group (No Intervention): Control group will receive contact referrals only. A referral includes a contact number to addiction treatment (primary care and/or specialty addiction care consistent with diagnostic criteria) and injury prevention services at the Yale Hospital Violence Intervention Program.

INTERVENTIONS:
Behavioral: Brief Negotiation Interview intervention (BNI) (adapted) — A brief motivational interview designed to increase motivation to reduce alcohol and/or cannabis use and engagement in treatment referral.
  Arms: Brief Negotiation Interview intervention (BNI) (adapted)

SUMMARY:
This study aims to improve a short motivational conversation to better help young adults who were injured in assaults and also use alcohol or cannabis. Researchers will gather both interview and survey data from young adults who came to the emergency department after an assault and currently use alcohol or cannabis. Guided by a theory about risky behaviors, the study will focus on how confident young people feel about making changes to their alcohol and cannabis use, and how their friends and family influence their alcohol and cannabis use and involvement in injuries from assault. The team will follow a step-by-step process used by the NIH to adapt and test the improved motivational conversation in the emergency department.

DETAILED DESCRIPTION:
Aim 1: Quantitatively and qualitatively assess self-efficacy, perceived peer and familial norms, and motivation to reduce alcohol and/or cannabis use and engage in treatment referral, among assault-injured emerging adults. AIM 2: Adapt the BNI for use among assault-injured emerging adults with alcohol and/or cannabis misuse in the ED. AIM 3: Determine the feasibility and acceptability of an adapted BNI among assault-injured emerging adults with alcohol and/or cannabis misuse presenting to the ED through a randomized pilot trial comparing those who have received the adapted BNI and treatment referrals to a referrals-only control group. The focus of this registration is the randomized pilot in Aim 3. Anticipated start dates will be reflected in the clinical trial component in Aim 3.

ELIGIBILITY:
Inclusion Criteria:

Aim 1:

* Be clients of the Yale Hospital Violence Intervention Program (YHVIP)
* Be between the ages of 18-25 y/o upon study enrollment
* Have sustained an intentional injury inflicted by another person not considered to be a boy/girlfriend, fiancée, or spouse in the past year
* Report current alcohol and/or cannabis misuse
* Be English-speaking and able to provide informed consent.

Aim 2 and 3:

* Present to Yale New Haven Hospital ED for an intentional injury inflicted by another person not considered to be a boy/girlfriend, fiancée, or spouse
* Be between the ages of 18-25 y/o upon study enrollment
* Report current alcohol and/or cannabis misuse
* Be English-speaking and able to provide informed consent.

Exclusion Criteria:

Aim 1:

* Be actively suicidal or severely cognitively impaired precluding informed consent
* Sustain an intentional injury from a boy/girlfriend, fiancée, or spouse or sexual assault
* Be incarcerated or in police custody
* Currently engaged in addiction treatment

Aim 2 and 3:

* Be actively suicidal or severely cognitively impaired precluding informed consent
* Sustain intentional injury from a boy/girlfriend, fiancée, spouse or by sexual assault
* Be incarcerated or in police custody
* Currently engaged in addiction treatment

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2026-08 (Estimated); Primary Completion 2028-02 (Estimated); Study Completion 2028-02 (Estimated)

PRIMARY OUTCOMES:
Feasibility assessed by recruitment | Day 0 and 30
  Recruitment measured as the percentage of those invited/those who enrolled
Feasibility assessed by randomization | Day 0 and 30
  Recruitment measured as the percentage of screened eligible participants who enroll/those who receive either intervention or control arm
Feasibility assessed by retention | Day 0 and 30
  Recruitment measured as the percentage of those enrolled who have received either intervention or control arm/ participants who have completed all 30-day follow up assessments
Acceptability assessed by Acceptability of Intervention Measure (AIM) | Day 0
  Acceptability of the intervention will be assessed using the Acceptability of Intervention Measure (AIM). It has 4-items scored on a 5-point Likert scale summed to achieve a total score. Total score range of 0-20. Higher scores indicate more acceptability.

CONTACTS AND LOCATIONS:
Overall Officials: Edouard Coupet, MD, MS, Principal Investigator — Yale University
Locations (1):
- Yale Department of Emergency Medicine, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual-level data will be shared 6 months after publication for up to 3 years